CLINICAL TRIAL: NCT00476398
Title: Evaluation of Patients With Non-cardiac Chest Pain Using PillCam Eso - a Wireless Imaging Capsule of the Esophagus.
Brief Title: Evaluation of Patients With Non-cardiac Chest Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Associate Physician, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2005P001321
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Non-Cardiac Chest Pain; Gastroesophageal Reflux Disease
Keywords: Capsule endoscopy; Wireless imaging; esophagus; stomach
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic capsule endoscopy (No Intervention): Patient with non-cardiac chest pain will undergo capsule endoscopy
  Interventions: Procedure: Capsule endoscopy

INTERVENTIONS:
Procedure: Capsule endoscopy — Patient will undergo a capsule endoscopy for the evaluation of their chest pain.

SUMMARY:
The purpose of this study is to find out how common diseases of the esophagus can cause chest pain. Gastroesophageal reflux disease (GERD), commonly known as heartburn, is a common cause of chest pain in patients that do not have heart problems. The study test is called PillCam Eso, it is a small, pill sized capsule that has a small camera inside it. The camera will take pictures of the esophagus and the stomach as it goes down. Findings of the PillCam Eso will be compared to findings during conventional upper endoscopy.

DETAILED DESCRIPTION:
Non-cardiac chest pain (NCCP) is defined by recurrent episodes of retrosternal chest pain in the absence of significant cardiovascular disease after a thorough cardiac evaluation. It accounts for 2-5% of all emergency department visits. Studies examining the prevalence of esophago-gastric lesions in patients with NCCP referred to gastroenterologists have found esophagitis, esophageal ulcers, hiatal hernias, gastritis, and gastric ulcers in 62% of patients. Advances in endoscopic technologies, particularly, the introduction of the wireless video-capsule (PillCam Eso) allows for the possibility of direct visualization of the upper gastrointestinal tract in the emergency department. During capsule endoscopy, a patient will swallow a pill-sized video-capsule, the wireless images of the gastrointestinal tract are transmitted to a computer. Findings of the PillCam Eso will be then compared to findings during conventional upper endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 80 years
* negative cardiac evaluation in the emergency department
* pre-established access to a primary care provider
* ability to give informed consent

Exclusion Criteria:

* known history of ischemic heart disease
* proton pump inhibitor therapy
* known or suspected obstructions or strictures in the gastrointestinal tract, including a history of Crohn's disease, gastrointestinal surgery other than cholecystectomy or appendectomy.
* permanent pacemakers/defibrillators or other implantable wireless devices
* known pregnancy
* unstable medical conditions
* inability to follow instructions
* active psychiatric conditions that preclude participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
endoscopy for evaluating the prevalence of esophago-gastric lesions in patients | 60 day

CONTACTS AND LOCATIONS:
Overall Officials: Julia J. Liu, MD, Principal Investigator — Brigham and Women's Hospital